CLINICAL TRIAL: NCT06369610
Title: Risk Stratified De-Escalated De-Intensified Treatment for High Risk Prostate Cancer Patients Based on Pathologic Criteria, Genetic Score, and Biologic Imaging
Brief Title: Risk Stratified De-escalated Hormone Therapy With Radiation Therapy for the Treatment of Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMROA2256; NCI-2024-03020 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-012591 (Other: Mayo Clinic Institutional Review Board); GMROA2256 (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2024-04-12; First posted 2024-04-17 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Oligometastatic Prostate Carcinoma; Prostate Adenocarcinoma
MeSH Terms: interventions — Abiraterone Acetate; Specimen Handling; Gonadotropin-Releasing Hormone; Magnetic Resonance Spectroscopy; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (radiation therapy) (Experimental): Patients undergo radiation therapy to the prostate bed over 2 - 6 weeks. Additionally, patients undergo PET, CT or MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy
- Group II (ADT, radiation therapy) (Experimental): Patients receive ADT SC or IM for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy to the prostate bed over 2 - 6 weeks starting on week 8-10 of ADT hormone therapy. Additionally, patients undergo PET, CT or MRI and blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Gonadotropin-releasing Hormone Analog; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy
- Group III (ADT, radiation therapy, abiraterone acetate) (Experimental): Patients receive ADT SC or IM with or without abiraterone acetate for up to 18 months in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy to identified areas over 2 - 6 weeks starting on week 8-10 of ADT hormone therapy. Additionally, patients undergo PET, CT or MRI and blood sample collection throughout the study.
  Interventions: Drug: Abiraterone Acetate; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Gonadotropin-releasing Hormone Analog; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Abiraterone Acetate — Given abiraterone acetate
  Other Names: BR9004; BR9004-1; CB7630; JNJ-212082; Yonsa; Zytiga
  Arms: Group III (ADT, radiation therapy, abiraterone acetate)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Gonadotropin-releasing Hormone Analog — Given SC or IM
  Other Names: GnRH Agonist; GnRH Analog; Gonadotropin-Releasing Hormone Agonist; Gonadotropin-Releasing Hormone Analogue; LH-RH agonist; LH-RH Analogs; LHRH Agonist; luteinizing hormone-releasing hormone agonist; Luteinizing Hormone-Releasing Hormone Analog
  Arms: Group II (ADT, radiation therapy); Group III (ADT, radiation therapy, abiraterone acetate)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase II trial tests how well risk based de-escalated hormone therapy (i.e., fewer treatments) with radiation works in treating patients with prostate cancer. Androgen deprivation therapy (ADT), such as gonadotropin-releasing hormone analogs (LHRH) and abiraterone acetate (Zytiga), lower the amount of the male hormone, testosterone, made by the body. This may help kill or stop the growth of tumor cells that need testosterone to grow. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill cancer cells and shrink tumors. Research has shown that long-term ADT is beneficial for patients with high-risk prostate cancer. However, there are few studies that determine ADT treatment based on risk factors. Giving risk based de-escalated ADT with radiation therapy may be as effective as giving more ADT in treating high-risk prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Recovery of the Expanded Prostate Cancer Index Composite (EPIC) hormonal domain to baseline levels at 2-years.

EXPLORATORY OBJECTIVES:

I. After completion of radiation therapy, determine the incidence of:

Ia. Grade 2 or greater genitourinary (GU) and gastrointestinal (GI) toxicity at 6 months (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0); Ib. Grade 3 or greater GU and GI toxicity at 6 months (CTCAE version 5.0); Ic. Patient-reported quality of life; Id. Impotence after the use of radiation therapy at 3 years; Ie. Freedom from biochemical failure (FFBF) at 5 years; If. Clinical failure: local and/or distant at 5 years; Ig. Salvage androgen deprivation use (SAD) at 5 years; Ih. Progression free survival: using clinical, biochemical and SAD as events at 5 years; Ij. Overall survival at 5 years; Ik. Disease-specific survival at 5 years. II. Determine overall GI and GU toxicity.

OUTLINE: Patients are assigned to 1 of 3 risk groups.

GROUP I (LOW RISK): Patients undergo radiation therapy to the prostate bed over 2 - 6 weeks.

GROUP II (INTERMEDIATE RISK): Patients receive ADT subcutaneously (SC) or intramuscularly (IM) for up to 12 months in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy to the prostate bed over 2 - 6 weeks starting on week 8-10 of ADT hormone therapy.

GROUP III: (HIGH RISK): Patients receive ADT SC or IM with or without abiraterone acetate for up to 18 months in the absence of disease progression or unacceptable toxicity. Patients also undergo radiation therapy to identified areas over 2 - 6 weeks starting on week 8-10 of ADT hormone therapy.

Additionally, patients undergo positron emission tomography (PET), computed tomography (CT) or magnetic resonance imaging (MRI), and blood sample collection throughout the trial.

After completion of study treatment, patients are followed up at months 3 and 12, then yearly for up to year 5 followed by every 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high risk prostate adenocarcinoma
* Pathologic stages T1c-T4, N0-Nx-N1, M0-1 as staged by the pathology report (AJCC Criteria 8th Edition [Ed].)
* One or more high risk features including Gleason 8-10, T3-T4, prostate specific antigen (PSA) ≥ 20
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must sign institutional review board (IRB) approved study specific informed consent
* Patients must complete all required pre-entry tests
* Patients must be at least 18 years old
* Oligometastatic prostate cancer defined as disease in up to 5 distant or regional areas (group 3 only)

Exclusion Criteria:

* Previous pelvic radiation
* Prior androgen suppression therapy for prostate cancer for more than 6 months
* Active rectal diverticulitis, Crohn's disease affecting the rectum or ulcerative colitis (non-active diverticulitis and Crohn's disease not affecting the rectum are allowed)
* Prior systemic chemotherapy for prostate cancer
* History of proximal urethral stricture requiring dilatation
* Current and continuing anticoagulation with warfarin sodium (Coumadin), heparin, low-molecular weight heparin, clopidogrel bisulfate (Plavix), or equivalent (unless it can be stopped to manage treatment related toxicity, to have a biopsy if needed, or place markers)
* Major medical, addictive or psychiatric illness which in the investigator's opinion, will prevent the consent process, completion of the treatment and/or interfere with follow-up. (Consent by legal authorized representative is not permitted for this study)
* Evidence of any other cancer within the past 5 years and < 50% probability of a 5 year survival. (Prior or concurrent diagnosis of basal cell or non-invasive squamous cell cancer of the skin is allowed)
* History of myocardial infarction or decompensated congestive heart failure (CHF) within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2027-04-22 (Estimated); Study Completion 2027-04-22 (Estimated)

PRIMARY OUTCOMES:
Hormonal domain scores | At baseline and up to 2 years
  Measured by the Expanded Prostate Cancer Index Composite. Comparison will be made using a one-sided, paired-difference t-test, with a Type I error rate of 0.025.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E. Vargas, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials